CLINICAL TRIAL: NCT05279378
Title: Correlation of Lung Ultrasonography With Chest CT Findings in Cancer Patients With COVID-19 Viral Pneumonia, an Observational Study
Brief Title: Correlation of Lung Ultrasonography With Chest CT Findings in Cancer Patients With COVID-19 Viral Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, salma zanaty rady, assistant lecturer, South Egypt Cancer Institute
Other Study IDs: IORG0006563
Record Dates: First submitted 2022-03-11; First posted 2022-03-15 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Cancer Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: lung ultrasonography versus CT — chest CT will be done before admission and LUS within first 24 h from admission into the quarantine sector. In addition to 2 weeks after admission.
  CT images will be reviewed by chest radiologist expert, who will calculate a CT severity score based on extension and distribution of GGOs and consolidations.
  All CT scans will be performed in supine position at end inspiration without intravenous administration of contrast media.
  Within 24 h from admission and CT scanning, bedside LUS will be performed by clinician who will be blind to chest CT findings.
  Examinations will be performed with the patient in the sitting position, systematically scanning the front and the back side of each hemithorax.
  Blood sample will be collected into 4 mL Vacuette containing EDTA. Samples will be stored on ice, processed within 30 min and plasma will be isolated by centrifugation at 2000g for 20 min at 4 °C. Plasma will be immediately frozen at - 80 °C in several aliquots.

SUMMARY:
Thoracic imaging, either with chest X-ray (CXR) or computed tomography (CT), is an essential part of the diagnosis of coronavirus disease-19 (COVID-19) in patients admitted to hospital with fever or respiratory symptoms.

Inspite of the results of PCR tests are the gold standard, the sensitivity of CT for diagnosing COVID-19 is 97%. The specific epidemic contingency makes CT an accurate tool to stratify patients based on imaging patterns, predicting poor outcomes and the need for ventilation.

Lung ultrasound (LUS) is widely used in emergency departments because it is broadly available, low-cost, and has a high accuracy for diagnosing pulmonary diseases.

Despite the diagnostic power of LUS and its influence on decision-making and therapeutic management, there are still significant barriers to the widespread use of this tool.

The advantages of LUS are more obvious in older patients with multimorbidity and restricted mobility, for whom high-quality CXR and CT scans are difficult to obtain. In the hands of experienced clinicians, LUS diagnostic accuracy for bacterial pneumonia is similar to chest CT.

However, a correlation between LUS and CT findings in patient urgently hospitalized for severe COVID-19 pneumonia remains to be determined.

COVID-19 leads to an aggressive inflammatory response that is actually the reaction of the immune system. Some patients exhibit pneumonia in both lungs, multi-organ failure, and even death. Individuals who have severe health conditions, like cancer, cardiovascular diseases, diabetes, and pulmonary diseases, are at higher risk of COVID-19 infection.

Also, this dysregulated immune response resulting in excessive production of inflammatory cytokines and chemokines (as IL-1ra, IL-6, IP-10, G-CSF, MCP-1, MIP-1α and TNF) causes the development of cytokine release syndrome (CRS) which is considered as pathologic underpinning for disease progression and lead to severe collateral tissue damage.

IL-6 may serve as a predictive biomarker for disease severity as its elevated levels were reported in several studies of COVID-19 infection. Also IL-6 levels were correlated with mortality in COVID-19 patients. IL-6 blockade is a promising strategy for COVID-induced CRS.

In particular, clinical epidemiological studies are needed to determine if IL-6 and/or other inflammatory cytokine levels predict subsequent development and persistence of long COVID 19 viral pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include cancer patients admitted to South Egypt Cancer Institute (SECI), Asyut University, Egypt with COVID-19 viral pneumonia in the period from March 2022 to December 2023, with ages ranging from 18 to 60 years old, of male or female gender, and CT Chest findings of CORAD 4, 5 and 6 with moderate and severe symptoms.
* All cancer patients are diagnosed COVID-19 by PCR from a nasopharyngeal swab.

Exclusion Criteria:

* Critical conditions need for ICU at the time of admission, presence of severe cardiorespiratory illness other than COVID-19 viral pneumonia, hepatic and renal diseases, coagulopathy, and patient refusal to share in our study will be considered as exclusion criteria.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cancer patients admitted to South Egypt Cancer Institute (SECI), Asyut University, Egypt with COVID-19 viral pneumonia in the period from March 2022 to December 2023, with ages ranging from 18 to 60 years old, of male or female gender, and CT Chest findings of CORAD 4, 5 and 6 with moderate and severe symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
comparing the CT versus LUS findings | 2 weeks
  comparing the CT versus LUS findings in cancer patients with moderate and severe COVID-19 viral pneumonia who will be admitted to our hospital and to correlate these findings with clinical features

SECONDARY OUTCOMES:
correlation of the results with the level of IL-6 | within 2 weeks
  correlate the results with the clinical data and laboratory data including the level of IL-6, D-dimer, serum ferritin and C-reactive protein (CRP) of those cancer patients during quarantine period.

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt cancei institute, Asyut, Egypt

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Sethuraman N, Jeremiah SS, Ryo A. Interpreting Diagnostic Tests for SARS-CoV-2. JAMA. 2020 Jun 9;323(22):2249-2251. doi: 10.1001/jama.2020.8259. No abstract available. PMID 32374370
- [Background] Kim H, Hong H, Yoon SH. Diagnostic Performance of CT and Reverse Transcriptase Polymerase Chain Reaction for Coronavirus Disease 2019: A Meta-Analysis. Radiology. 2020 Sep;296(3):E145-E155. doi: 10.1148/radiol.2020201343. Epub 2020 Apr 17. PMID 32301646
- [Background] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Background] Colombi D, Bodini FC, Petrini M, Maffi G, Morelli N, Milanese G, Silva M, Sverzellati N, Michieletti E. Well-aerated Lung on Admitting Chest CT to Predict Adverse Outcome in COVID-19 Pneumonia. Radiology. 2020 Aug;296(2):E86-E96. doi: 10.1148/radiol.2020201433. Epub 2020 Apr 17. PMID 32301647
- [Background] Kwee TC, Kwee RM. Chest CT in COVID-19: What the Radiologist Needs to Know. Radiographics. 2020 Nov-Dec;40(7):1848-1865. doi: 10.1148/rg.2020200159. Epub 2020 Oct 23. PMID 33095680
- [Background] Gargani L, Picano E. The risk of cumulative radiation exposure in chest imaging and the advantage of bedside ultrasound. Crit Ultrasound J. 2015 Mar 28;7:4. doi: 10.1186/s13089-015-0020-x. eCollection 2015. PMID 25883779
- [Background] Mossa-Basha M, Meltzer CC, Kim DC, Tuite MJ, Kolli KP, Tan BS. Radiology Department Preparedness for COVID-19: Radiology Scientific Expert Review Panel. Radiology. 2020 Aug;296(2):E106-E112. doi: 10.1148/radiol.2020200988. Epub 2020 Mar 16. No abstract available. PMID 32175814
- [Background] de Alencar JCG, Marchini JFM, Marino LO, da Costa Ribeiro SC, Bueno CG, da Cunha VP, Lazar Neto F, Brandao Neto RA, Souza HP; COVID U. S. P. Registry Team. Lung ultrasound score predicts outcomes in COVID-19 patients admitted to the emergency department. Ann Intensive Care. 2021 Jan 11;11(1):6. doi: 10.1186/s13613-020-00799-w. PMID 33427998
- [Background] Georgopoulos D, Xirouchaki N, Volpicelli G. Lung ultrasound in the intensive care unit: let's move forward. Intensive Care Med. 2014 Oct;40(10):1592-4. doi: 10.1007/s00134-014-3484-4. Epub 2014 Sep 18. No abstract available. PMID 25231292
- [Background] Nouvenne A, Zani MD, Milanese G, Parise A, Baciarello M, Bignami EG, Odone A, Sverzellati N, Meschi T, Ticinesi A. Lung Ultrasound in COVID-19 Pneumonia: Correlations with Chest CT on Hospital admission. Respiration. 2020;99(7):617-624. doi: 10.1159/000509223. Epub 2020 Jun 22. PMID 32570265
- [Background] Ticinesi A, Scarlata S, Nouvenne A, Lauretani F, Incalzi RA, Ungar A; GRETA (Gruppo di Ricerca sull'Ecografia Toracica nell'Anziano) Group of the Italian Society of Gerontology and Geriatrics (SIGG). The Geriatric Patient: The Ideal One for Chest Ultrasonography? A Review From the Chest Ultrasound in the Elderly Study Group (GRETA) of the Italian Society of Gerontology and Geriatrics (SIGG). J Am Med Dir Assoc. 2020 Apr;21(4):447-454.e6. doi: 10.1016/j.jamda.2019.06.018. Epub 2019 Aug 6. PMID 31399360
- [Background] Berlet T. Thoracic ultrasound for the diagnosis of pneumonia in adults: a meta-analysis. Respir Res. 2015 Jul 25;16(1):89. doi: 10.1186/s12931-015-0248-9. No abstract available. PMID 26205975
- [Background] Fu Y, Cheng Y, Wu Y. Understanding SARS-CoV-2-Mediated Inflammatory Responses: From Mechanisms to Potential Therapeutic Tools. Virol Sin. 2020 Jun;35(3):266-271. doi: 10.1007/s12250-020-00207-4. Epub 2020 Mar 3. PMID 32125642
- [Background] Liu F, Zhang Q, Huang C, Shi C, Wang L, Shi N, Fang C, Shan F, Mei X, Shi J, Song F, Yang Z, Ding Z, Su X, Lu H, Zhu T, Zhang Z, Shi L, Shi Y. CT quantification of pneumonia lesions in early days predicts progression to severe illness in a cohort of COVID-19 patients. Theranostics. 2020 Apr 27;10(12):5613-5622. doi: 10.7150/thno.45985. eCollection 2020. PMID 32373235
- [Background] Nishiga M, Wang DW, Han Y, Lewis DB, Wu JC. COVID-19 and cardiovascular disease: from basic mechanisms to clinical perspectives. Nat Rev Cardiol. 2020 Sep;17(9):543-558. doi: 10.1038/s41569-020-0413-9. Epub 2020 Jul 20. PMID 32690910
- [Background] Dai M, Liu D, Liu M, Zhou F, Li G, Chen Z, Zhang Z, You H, Wu M, Zheng Q, Xiong Y, Xiong H, Wang C, Chen C, Xiong F, Zhang Y, Peng Y, Ge S, Zhen B, Yu T, Wang L, Wang H, Liu Y, Chen Y, Mei J, Gao X, Li Z, Gan L, He C, Li Z, Shi Y, Qi Y, Yang J, Tenen DG, Chai L, Mucci LA, Santillana M, Cai H. Patients with Cancer Appear More Vulnerable to SARS-CoV-2: A Multicenter Study during the COVID-19 Outbreak. Cancer Discov. 2020 Jun;10(6):783-791. doi: 10.1158/2159-8290.CD-20-0422. Epub 2020 Apr 28. PMID 32345594
- [Background] Yue H, Bai X, Wang J, Yu Q, Liu W, Pu J, Wang X, Hu J, Xu D, Li X, Kang N, Li L, Lu W, Feng T, Ding L, Li X, Qi X; Gansu Provincial Medical Treatment Expert Group of COVID-19. Clinical characteristics of coronavirus disease 2019 in Gansu province, China. Ann Palliat Med. 2020 Jul;9(4):1404-1412. doi: 10.21037/apm-20-887. Epub 2020 Jul 13. PMID 32692208
- [Background] Parsons PE, Eisner MD, Thompson BT, Matthay MA, Ancukiewicz M, Bernard GR, Wheeler AP; NHLBI Acute Respiratory Distress Syndrome Clinical Trials Network. Lower tidal volume ventilation and plasma cytokine markers of inflammation in patients with acute lung injury. Crit Care Med. 2005 Jan;33(1):1-6; discussion 230-2. doi: 10.1097/01.ccm.0000149854.61192.dc. PMID 15644641
- [Background] Giamarellos-Bourboulis EJ, Netea MG, Rovina N, Akinosoglou K, Antoniadou A, Antonakos N, Damoraki G, Gkavogianni T, Adami ME, Katsaounou P, Ntaganou M, Kyriakopoulou M, Dimopoulos G, Koutsodimitropoulos I, Velissaris D, Koufargyris P, Karageorgos A, Katrini K, Lekakis V, Lupse M, Kotsaki A, Renieris G, Theodoulou D, Panou V, Koukaki E, Koulouris N, Gogos C, Koutsoukou A. Complex Immune Dysregulation in COVID-19 Patients with Severe Respiratory Failure. Cell Host Microbe. 2020 Jun 10;27(6):992-1000.e3. doi: 10.1016/j.chom.2020.04.009. Epub 2020 Apr 21. PMID 32320677
- [Background] Patrucco F, Albera C, Bellocchia M, Foci V, Gavelli F, Castello LM, Bellan M, Sainaghi PP, Airoldi C, Balbo PE, Solidoro P. SARS-CoV-2 Detection on Bronchoalveolar Lavage: An Italian Multicenter experience. Respiration. 2020;99(11):970-978. doi: 10.1159/000511964. Epub 2020 Oct 19. PMID 33075793
- [Background] Wasilewski PG, Mruk B, Mazur S, Poltorak-Szymczak G, Sklinda K, Walecki J. COVID-19 severity scoring systems in radiological imaging - a review. Pol J Radiol. 2020 Jul 17;85:e361-e368. doi: 10.5114/pjr.2020.98009. eCollection 2020. PMID 32817769
- [Background] Falster C, Jacobsen N, Wulff Madsen L, Dahlerup Rasmussen L, Davidsen JR, Christie Knudtzen F, Nielsen SL, Johansen IS, Laursen CB. Lung ultrasound may be a valuable aid in decision making for patients admitted with COVID-19 disease. Eur Clin Respir J. 2021 Apr 7;8(1):1909521. doi: 10.1080/20018525.2021.1909521. PMID 33889342
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Proposal for International Standardization of the Use of Lung Ultrasound for Patients With COVID-19: A Simple, Quantitative, Reproducible Method. J Ultrasound Med. 2020 Jul;39(7):1413-1419. doi: 10.1002/jum.15285. Epub 2020 Apr 13. PMID 32227492
- See also: Diagnostic Performance of CT and Reverse Transcriptase Polymerase Chain Reaction for Coronavirus Disease 2019: A Meta-Analysis — https://pubmed.ncbi.nlm.nih.gov/32301646/
- See also: Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases — https://pubmed.ncbi.nlm.nih.gov/32101510/
- See also: Well-aerated Lung on Admitting Chest CT to Predict Adverse Outcome in COVID-19 Pneumonia. — https://pubmed.ncbi.nlm.nih.gov/32301647/
- See also: The risk of cumulative radiation exposure in chest imaging and the advantage of bedside ultrasound — https://pubmed.ncbi.nlm.nih.gov/25883779/
- See also: The risk of cumulative radiation exposure in chest imaging and the advantage of bedside ultrasound — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4392040/
- See also: Lung ultrasound score predicts outcomes in COVID-19 patients admitted to the emergency department — https://pubmed.ncbi.nlm.nih.gov/33427998/
- See also: Lung ultrasound in the intensive care unit: let's move forward — https://pubmed.ncbi.nlm.nih.gov/25231292/
- See also: Lung Ultrasound in COVID-19 Pneumonia: Correlations with Chest CT on Hospital admission — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7360505/
- See also: The Geriatric Patient: The Ideal One for Chest Ultrasonography? A Review From the Chest Ultrasound in the Elderly Study Group (GRETA) of the Italian Society of Gerontology and Geriatrics (SIGG) — https://pubmed.ncbi.nlm.nih.gov/31399360/
- See also: Thoracic ultrasound for the diagnosis of pneumonia in adults: A meta-analysis — https://pubmed.ncbi.nlm.nih.gov/28099332/
- See also: Understanding SARS-CoV-2-Mediated Inflammatory Responses: From Mechanisms to Potential Therapeutic Tools — https://pubmed.ncbi.nlm.nih.gov/32125642/
- See also: CT quantification of pneumonia lesions in early days predicts progression to severe illness in a cohort of COVID-19 patients — https://pubmed.ncbi.nlm.nih.gov/32345594/
- See also: COVID-19 and cardiovascular disease: from basic mechanisms to clinical perspectives — https://pubmed.ncbi.nlm.nih.gov/32692208/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15644641/
- See also: Patients with Cancer Appear More Vulnerable to SARS-CoV-2: A Multicenter Study during the COVID-19 Outbreak — https://pubmed.ncbi.nlm.nih.gov/32320677/
- See also: Clinical characteristics of coronavirus disease 2019 in Gansu province — https://pubmed.ncbi.nlm.nih.gov/33075793/
- See also: Lung ultrasound score predicts outcomes in COVID-19 patients admitted to the emergency department. — https://pubmed.ncbi.nlm.nih.gov/32817769/
- See also: Lung ultrasound in the intensive care unit: let's move forward — https://pubmed.ncbi.nlm.nih.gov/33889342/
- See also: Lung Ultrasound in COVID-19 Pneumonia: Correlations with Chest CT on Hospital admission — https://pubmed.ncbi.nlm.nih.gov/32227492/